CLINICAL TRIAL: NCT00315133
Title: Autologous Hematopoietic Stem Cell Transplantation for Early Onset Type 1 Diabetes Mellitus- a Phase I/II Study
Brief Title: Safety and Efficacy Study of Autologous Stem Cell Transplantation for Early Onset Type I Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Northwestern University (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Julio C. Voltarelli, Julio C. Voltarelli, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCFMRPUSP
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes mellitus; Stem cells; Autologous stem cell transplantation; Autoimmune diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases | interventions — Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant arm (Experimental): This is a single arm study. The intervention is immunosuppression and autologous stem cell transplantation.
  Interventions: Procedure: Immunosuppression and autologous stem cell transplantation

INTERVENTIONS:
Procedure: Immunosuppression and autologous stem cell transplantation — Immunosuppression and autologous stem cell transplantation: Mobilization of hematopoietic stem cells (HSC) with cyclophosphamide (2 g/m2) and granulocyte-colony stimulating factor (G-CSF, 10 ug/kg/d), followed by collection and cryopreservation of unselected HSC and conditioning with cyclophosphamide (200 mg/kg) plus rabbit anti-thymocyte globulin (ATG 4.5 mg/kg).

SUMMARY:
The study evaluates the effect of inactivation of the immune system with chemotherapy and immunotherapy and infusion of bone marrow stem cells in early onset type 1 diabetes mellitus. We hypothesize that reprograming the immune system will stop immune aggression to the insulin producing cells allowing their regeneration and thus decreasing or eliminating the need of exogenous insulin.

DETAILED DESCRIPTION:
Patients from 12 to 35 years old with type I diabetes mellitus proved by anti-pancreatic beta cell antibodies and recently diagnosed (less than 6 weeks) will be included in this study. Peripheral blood hematopoietic stem cells will be mobilized from bone marrow of the patient with cyclophosphamide plus G-CSF (granulocyte-colony stimulating factor), collected by leukapheresis and cryopreserved. After 2-3 weeks, high dose immunosuppression is given (cyclophosphamide 200 mg/kg plus rabbit antithymocyte globulin 4.5 mg/kg) and stem cells are thawed and injected intravenously. This procedure is performed in isolated rooms at the Bone Marrow Transplantation Unit of the School of Medicine of Ribeirão Preto, University of São Paulo, Brazil. Patients are discharged from the hospital after engraftment and closely followed up to 2 months after transplantation (with at least weekly outpatient visits) and continue the followup for 5 years after transplantation. Clinical, hematological, metabolical and immunological evaluations are performed to analyse the effect of the transplant in the disease and in the hematopoetic and immunologic systems of the body. Patients fitting the inclusion criteria but not agreeing to perform the transplantation are the control group and they will be followed in parallel with transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus diagnosed by clinical/metabolic parameters and positive anti-GAD antibodies
* Less than 12 weeks from diagnosis

Exclusion Criteria:

* Previous diabetic ketoacidosis
* Pregnancy
* Severe psychiatric disorder
* Severe organic impairment (renal, hepatic, cardiac, pulmonary)
* Active infectious disease
* Previous or present neoplastic disease

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2003-12; Primary Completion 2010-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
C-peptide levels | Every 6 months
  Stimulated C-peptide levels will be measured.

SECONDARY OUTCOMES:
Transplant-related toxicity | Every 6 months or when reported
Anti-GAD titres | Every 6 months
Exogenous insulin dose | Every 6 months
  Number of international insulin units per kilogram per day in use will be registered.
Hemoglobin A1C | Every 6 months
  Hb A1C will be measured.
Immunologic reconstitution parameters | Yearly
Quality of Life | Every year
  SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Julio C Voltarelli, MD PhD, Principal Investigator — University Hospital, School of Medicine of Ribeirão Preto, Brazil; Maria C Oliveira, MD PhD, Study Chair — University Hospital, Ribeirão Preto Medical School, Brazil
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, Ribeirão Preto, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared if the responsible investigators feel it may increase understanding, reliability and reproducibility of the present study.

REFERENCES:
- [Background] Burt RK, Oyama Y, Traynor A, Kenyon NS. Hematopoietic stem cell therapy for type 1 diabetes: induction of tolerance and islet cell neogenesis. Autoimmun Rev. 2002 May;1(3):133-8. doi: 10.1016/s1568-9972(02)00033-2. PMID 12849006
- [Result] Voltarelli JC, Couri CE, Stracieri AB, Oliveira MC, Moraes DA, Pieroni F, Coutinho M, Malmegrim KC, Foss-Freitas MC, Simoes BP, Foss MC, Squiers E, Burt RK. Autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2007 Apr 11;297(14):1568-76. doi: 10.1001/jama.297.14.1568. PMID 17426276
- [Result] Couri CE, Oliveira MC, Stracieri AB, Moraes DA, Pieroni F, Barros GM, Madeira MI, Malmegrim KC, Foss-Freitas MC, Simoes BP, Martinez EZ, Foss MC, Burt RK, Voltarelli JC. C-peptide levels and insulin independence following autologous nonmyeloablative hematopoietic stem cell transplantation in newly diagnosed type 1 diabetes mellitus. JAMA. 2009 Apr 15;301(15):1573-9. doi: 10.1001/jama.2009.470. PMID 19366777